CLINICAL TRIAL: NCT04911790
Title: Safety Observation of the Inactivated SARS-CoV-2 Vaccine (Vero Cell) in Population Aged 18 Years and Older: A Multicenter,Open-label Study
Brief Title: Safety of an Inactivated SARS-CoV-2 Vaccine for Prevention of COVID-19 in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4002
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Participant will receive two doses inactivated SARS-CoV-2 vaccine . Vaccine will given by intramuscular injection on day 0 and day 28.
  Interventions: Biological: Experimental Group

INTERVENTIONS:
Biological: Experimental Group — SARS-CoV-2 Inactivated Vaccine 600SU inactivated virus in 0·5 mL of aluminiumhydroxide solution per injection
  Other Names: CoronaVac

SUMMARY:
This study is a multi-center and open design, phase Ⅳ clinical trial of an inactivated SARS-CoV-2 vaccine (CoronaVac) manufactured by Sinovac Research and Development Co., Ltd.The purpose of this study is to evaluate the safety of the SARS-CoV-2 Inactivated vaccine in population aged 18 years years and older and in people with pre-existing disease to provide reference for improving the immunization strategy of COVID-19 vaccine.

DETAILED DESCRIPTION:
This study is a multi-center and open design, phase Ⅳ clinical trial in population aged 18 years years and older. The experimental vaccine will be manufactured by Sinovac Research and Development Co.,Ltd.The study is planned to be carried out in 11 provinces from May 2021 to December 2022, including Liaoning, Heilongjiang, Anhui, Fujian, Jiangxi, Hubei, Guangxi, Chongqing, Guizhou, Yunnan and Gansu. Each province will serve as a research center, and each research center will select the corresponding research site.A total of 121000 subjects will be enrolled with11000 for each research center, including at least 2000 people with pre-existing disease and at least 4000 people in the elderly group (60 years old and above) (including patients with pre-existing disease).And subjects will receive two doses of vaccine on day 0 and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Have not received any COVID-19 vaccine in the past or at least one dose of CoronaVac manufactured by Sinovac Research and Development Co.,Ltd;
* Population aged 18 years and above;
* The subjects can understand and voluntarily sign the informed consent form and participate in the follow-up;

Exclusion Criteria:

* History of severe allergy to the vaccine such as acute allergic reaction,angioedema and dyspnea ;
* Severe neurological disease such as transverse myeliti,Guillain-Barre Syndrome and demyelinating disorders;
* Acute diseas,acute onset of chronic disease and severe chronic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131650 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-7 after each dose vaccination
  Incidence rate of adverse reactions within 0~7 days after each dose in all populations.

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-7 after each dose vaccination
  Incidence of adverse reactions within 0~7 days after each dose in the population with pre-existing disease.
Safety index-incidence of adverse reactions | Day 0-28 after each dose vaccination
  Incidence rate of adverse reactions within 0~28 days after each dose in all populations.
Safety index-incidence of adverse reactions | Day 0-28 after each dose vaccination
  Incidence of adverse reactions within 0~28 days after each dose in the population with pre-existing disease.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Liu, Doctor, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention; Xing Fang, Principal Investigator — Liaoning Provincial Center for Disease Control and Prevention; Zhaodan Sun, Principal Investigator — HeilongjiangProvincial Center for Disease Control and Prevention; Fubing Wang, Principal Investigator — Hefei Provincial Center for Disease Control and Prevention; Dongjuan Zhang, Principal Investigator — Center for Disease Control and Prevention, Fujian; Shicheng Guo, Principal Investigator — Jiangxi Provincial Center for Disease Control and Prevention; Yeqing Tong, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention; Qiuyun Deng, Principal Investigator — Guangxi Center for Disease Control and Prevention; Qing Wang, Principal Investigator — Chongqing Center for Disease Control and Prevention; Ruizhi Zhang, Principal Investigator — Guizhou Provincial Center for Disease Control and Prevention; Xiaoshu Zhang, Principal Investigator — Gansu Provincial Center for Disease Control and Prevention
Locations (1):
- Yongping Center for Diseases Control and Prevention, Dali, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang H, Li Z, Zhang R, Guo S, Wang B, Fang X, Zhang D, Zhang X, Tong Y, Wang Q, Deng Q, Sun Z, Liu X, Gao Y. Safety of primary immunization using inactivated SARS-CoV-2 vaccine (CoronaVac(R)) among population aged 3 years and older in a large-scale use: A multi-center open-label study in China. Vaccine. 2023 Feb 10;41(7):1354-1361. doi: 10.1016/j.vaccine.2023.01.020. Epub 2023 Jan 13. PMID 36658045